CLINICAL TRIAL: NCT00634465
Title: A Biomechanical Assessment of the AST Stabilimax BAR Using Radiostereometric Analysis (RSA)
Status: Withdrawn | Type: Observational
Why Stopped: low enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Nathaniel Ordway, Orthopedic Surgery
Other Study IDs: Stabilimax Bar
Record Dates: First submitted 2008-03-04; First posted 2008-03-13 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Assess Motion in Flexion/Extension and Lateral Bending of the Lumbar Vertebrae in Vivo Following Motion Sparing Surgery Using Radiostereometric Analysis (RSA.)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Device: RSA Beads

INTERVENTIONS:
Device: RSA Beads — Radiostereometric Analysis, or RSA, is an accurate in vivo measurement technique using two simultaneous radiographs. It provides researchers with three dimensional motion analyses to look not only at routine flexion/extension, but also other rotational and translational changes

SUMMARY:
Assessment of segmental spine motion has been and continues to be, a difficult clinical problem. Errors of up to 10 degrees for simple measurements of flexion, extension and side bending have been recorded using conventional radiographs (xrays.) These errors are usually associated with the inability to acquire three-dimensional positions and inaccurate reference points. It has, therefore, been extremely difficult to measure small changes in vertebral alignment, which may prove to be an early, clinically significant, indicator of potential problems. Radiostereometric Analysis, or RSA, is an accurate in vivo measurement technique using two simultaneous radiographs. It provides researchers with three dimensional motion analyses to look not only at routine flexion/extension, but also other rotational and translational changes. The measurement accuracy offered by this technique far exceeds the manual techniques currently used. The purpose of this study is to assess the amount of motion in the lumbar spine in patients with the AST Stabilimax BAR. The AST Stabilimax BAR is designed to allow for motion in the spine while providing the necessary stability to the spinal segment. The amount and degree of this motion is currently unknown clinically. By using tantalum bead markers placed in the spine at the time of the surgery, RSA analysis can determine the amount and degree of motion of the implanted construct. Two questions will be examined with this data: 1) what is the amount of sagittal and coronal plane motion that occurs in vivo with the AST Stabilimax BAR system? and 2) will this change over the 2 year time frame for this study?

DETAILED DESCRIPTION:
Radiostereometric Analysis, or RSA, is an accurate in vivo measurement technique using two simultaneous radiographs. It provides researchers with three dimensional motion analyses to look not only at routine flexion/extension, but also other rotational and translational changes. The measurement accuracy offered by this technique far exceeds the manual techniques currently used. Utilization of the RSA technology at the IHP and the United States is in its infancy. The investigators have placed much effort over the past 2-3 years to put the necessary dedicated resources and personnel in place. This has been a collaborative effort between the Department of Orthopedic Surgery and the Imaging Core at IHP. Preliminary work on the accuracy, reliability, and surgical planning for use of RSA has been completed and presented at national conferences.

The purpose of this study is to assess the amount of motion in the lumbar spine in patients with the AST Stabilimax BAR. The AST Stabilimax BAR is designed to allow for motion in the spine while providing the necessary stability to the spinal segment. The amount and degree of this motion is currently unknown clinically, but has been biomechanically tested in vitro. By using tantalum bead markers placed in the spine at the time of the surgery, RSA analysis can determine the amount and degree of motion the implant provides. Two questions will be examined with this data: 1) what is the amount of sagittal and coronal plane motion that occurs in vivo with the AST Stabilimax BAR system? and 2) will this change over the 2 year time frame for this study?

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled to have lumbar surgery to receive the AST Stabilimax BAR
* All subjects must be skeletally mature, between the ages of 18-75

Exclusion Criteria:

* Pregnant women will be excluded due to added radiation exposure
* Prisoners will also be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center, non-randomized study. 10 Subjects who are identified to receive the AST Stabilimax BAR device will be approached to participate in this study. All subjects will receive 10 RSA tantalum beads (5 in each vertebra) at the time of their lumbar surgery. After surgery, subjects will have the biplanar xrays taken. The biplanar xrays will be taken from 5 standing positions: neutral, flexion (bending forward), extension (bending backwards), left side bending, and right side bending. RSA analysis will be completed to determine the amount of motion on sagittal and coronal planes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States